CLINICAL TRIAL: NCT02726308
Title: Dexamethasone Alone Versus in Combination With Intra-operative Super-hydration for Prevention of Postoperative Nausea and Vomiting in Female Patients Undergoing Laparoscopic Cholecystectomy: A Randomized Clinical Trial
Brief Title: Dexamethasone With Super-hydration for Prevention of Postoperative Nausea and Vomiting
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sayed Kaoud Abd-Elshafy, Associate Professor (Anesthesiology and Critical Care)- College of Medicine-Assiut University, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB0000871550
Record Dates: First submitted 2016-03-29; First posted 2016-04-01 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Nausea and Vomiting, Postoperative
Keywords: Dexamethasone; Super-hydration; Laparoscopic Cholecystectomy; Nausea; Vomiting; Postoperative
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Nausea; Vomiting | interventions — Dexamethasone; Calcium Dobesilate; Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexamethasone Group (Active Comparator): I.V. Dexamethasone 5 mg just before induction plus intra-operative 10 ml/kg Ringer's lactate solution.
  Interventions: Drug: Dexamethasone; Drug: 10 ml/kg Ringer's lactate
- Dexamethasone and super-hydration Group (Active Comparator): I.V. Dexamethasone 5 mg just before induction of anesthesia plus intraoperative 30 ml/kg Ringer's lactate solution
  Interventions: Drug: Dexamethasone; Drug: 30 ml/kg Ringer's lactate

INTERVENTIONS:
Drug: Dexamethasone — 5 mg I.V. Dexamethasone just before induction
  Other Names: Decadron
Drug: 10 ml/kg Ringer's lactate — Intra-operative 10 ml/kg Ringer's lactate solution .
  Other Names: Normal hydration
  Arms: Dexamethasone Group
Drug: 30 ml/kg Ringer's lactate — Intra-operative 30 ml/kg Ringer's lactate solution .
  Other Names: super-hydration
  Arms: Dexamethasone and super-hydration Group

SUMMARY:
Postoperative nausea and vomiting (PONV) are the most common and distressing side effects following Laparoscopic cholecystectomy

DETAILED DESCRIPTION:
In the operating room, standard monitors included electrocardiogram, noninvasive arterial blood pressure, arterial oxygen saturation, and end-tidal carbon dioxide were connected. All patients received standardized anesthetic technique. At the end of surgery, gastric contents were suctioned via an orogastric tube before extubation. Atropine and neostigmine (1/2.5 mg) was given slowly I.V. to antagonize the residual neuromuscular block. Then, the trachea was extubated. Then, patients were transferred to the post-anesthesia care unit in a stable condition. Patients were allowed to drink liquids as soon as requested.

ELIGIBILITY:
Inclusion Criteria:

American Society of Anesthesiologists (ASA) physical status I or II aged Elective laparoscopic cholecystectomy

Exclusion Criteria:

Steroids use within the last 3 days before surgery Antiemetic use within the last 3 days before surgery Opioids use within the last 3 days before surgery. Patients with liver, cardiac or renal diseases Patients with Pregnancy Patients with Bmi ˃ 30kg/m2 Patients with Delayed wound healing Open surgery

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2015-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Postoperative Nausea and Vomiting (PONV) | Within the first 24 hours postoperatively
  A nurse, who was unaware about the groups to which the patient belonged, evaluated patients at 0, 6, and 24 h after surgery for any symptoms of nausea, retching, or vomiting. PONV is classified as early, if occurring up to 6h after surgery, or late, if occurring between 6 h up to 24 postoperatively.
  A Verbal Descriptive Scale (VDS), was used to assess the severity of PONV: no PONV (grade 0), mild PONV (grade 1), moderate PONV (grade 2) and severe PONV (grade 3)

SECONDARY OUTCOMES:
Total number of patients who had nausea, vomiting or retching | Within the first 24 hours postoperatively
  Total number of patients who had nausea, vomiting or retching (number)
Antiemetic usage | Within the first 24 hours postoperatively
  Total amount of ondansetron consumption (mg)
Pain Score | Within the first 24 hours postoperatively
  A visual analogue scale (appropriate score)
Total analgesic consumption | Within the first 24 hours postoperatively
  I.V Pethidine (mg)
Incidence of wound infection | Within the first week postoperatively
  Number of patients
Incidence of delayed wound healing | Within the first week postoperatively
  Number of patients

CONTACTS AND LOCATIONS:
Overall Officials: sayed abd elshafy, MD, Principal Investigator — associate professor of anesthesia and critical care
Locations (1):
- Faculty of Medicine, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided